CLINICAL TRIAL: NCT05344417
Title: Impact of Low Pressure Pneumoperitoneum on Postoperative Ileus and Gastrointestinal Dysfunction in Patients Undergoing Laparoscopic Large Bowel Surgery
Brief Title: Low Pressure Pneumoperitoneum and Postoperative Ileus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Fedias Christofi, Professor and Vice Chair of Research, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021H0262
Record Dates: First submitted 2022-03-31; First posted 2022-04-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Ileus; Gastrointestinal Dysfunction
MeSH Terms: interventions — Neuromuscular Blockade

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Arm 1: Standard of Care (No Intervention): 25 patients undergoing laparoscopic right hemi-colectomies or sigmoid resections using high pneumoperitoneum pressure with conventional insufflation under moderate neuromuscular blockade with rocuronium and neuromuscular blockade reversal with neostigmine. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.
- Arm 2A: Conventional Pneumoperitoneum and Moderate Blockade (Experimental): 25 patients undergoing laparoscopic right hemi-colectomies or sigmoid resections using high pneumoperitoneum pressure with conventional insufflation under moderate neuromuscular blockade with rocuronium and neuromuscular blockade reversal with sugammadex. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.
  Interventions: Procedure: Pneumoperitoneum Pressure; Procedure: Neuromuscular blockade; Device: Pneumoperitoneum insufflation device; Drug: Neuromuscular blockade reversal
- Arm 2B: AirSeal® Pneumoperitoneum and Moderate Blockade (Experimental): 25 patients undergoing laparoscopic right hemi-colectomies or sigmoid resections using high pneumoperitoneum pressure with AirSeal® trademark (TM) system under moderate neuromuscular blockade with rocuronium and neuromuscular blockade reversal with sugammadex. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.
  Interventions: Procedure: Pneumoperitoneum Pressure; Procedure: Neuromuscular blockade; Device: Pneumoperitoneum insufflation device; Drug: Neuromuscular blockade reversal
- Arm 3A: Conventional Pneumoperitoneum and Deep Blockade (Experimental): 25 patients undergoing laparoscopic right hemi-colectomies or sigmoid resections using low pneumoperitoneum pressure with conventional insufflation under deep neuromuscular blockade with rocuronium and neuromuscular blockade reversal with sugammadex. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.
  Interventions: Procedure: Pneumoperitoneum Pressure; Procedure: Neuromuscular blockade; Device: Pneumoperitoneum insufflation device; Drug: Neuromuscular blockade reversal
- Arm 3B: AirSeal® Pneumoperitoneum and Deep Blockade (Experimental): 25 patients undergoing laparoscopic right hemi-colectomies or sigmoid resections using low pneumoperitoneum pressure with AirSeal® TM system under deep neuromuscular blockade with rocuronium and neuromuscular blockade reversal with sugammadex. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.
  Interventions: Procedure: Pneumoperitoneum Pressure; Procedure: Neuromuscular blockade; Device: Pneumoperitoneum insufflation device; Drug: Neuromuscular blockade reversal

INTERVENTIONS:
Procedure: Pneumoperitoneum Pressure — Low Pneumoperitoneum Pressure: defined as an intrabdominal pressure between 8-12 mmHg during the laparoscopic procedure.
  High Pneumoperitoneum pressure: defined as an intrabdominal pressure of 15 mmHg or more during the laparoscopic procedure.
  Note: surgeons will set the pneumoperitoneum at the lowest value they are comfortable with based on their surgical criteria
  Arms: Arm 2A: Conventional Pneumoperitoneum and Moderate Blockade; Arm 2B: AirSeal® Pneumoperitoneum and Moderate Blockade; Arm 3A: Conventional Pneumoperitoneum and Deep Blockade; Arm 3B: AirSeal® Pneumoperitoneum and Deep Blockade
Procedure: Neuromuscular blockade — Moderate neuromuscular blockade: defined as the presence of 1 or 2 responses after train-of-four stimulation.
  Deep neuromuscular blockade: defined as no response to train-of-four stimulation and 1 or less responses after post-tetanic count stimulation.
  Arms: Arm 2A: Conventional Pneumoperitoneum and Moderate Blockade; Arm 2B: AirSeal® Pneumoperitoneum and Moderate Blockade; Arm 3A: Conventional Pneumoperitoneum and Deep Blockade; Arm 3B: AirSeal® Pneumoperitoneum and Deep Blockade
Device: Pneumoperitoneum insufflation device — AirSeal® device or Olympus "standard of care" insufflation device. Both devices are approved for use in laparoscopic gastrointestinal surgeries.
  Arms: Arm 2A: Conventional Pneumoperitoneum and Moderate Blockade; Arm 2B: AirSeal® Pneumoperitoneum and Moderate Blockade; Arm 3A: Conventional Pneumoperitoneum and Deep Blockade; Arm 3B: AirSeal® Pneumoperitoneum and Deep Blockade
Drug: Neuromuscular blockade reversal — Neostigmine: for Arm 1 only (standard use).
  Sugammadex: will be used for the other arms in the study.
  All drugs used in our randomized trial (neuromuscular blockade with rocuronium and reversal with neostigmine or sugammadex) are standard of care and approved for use by our institutional Institutional Review Board (IRB) Ethics Committee for this trial.
  Arms: Arm 2A: Conventional Pneumoperitoneum and Moderate Blockade; Arm 2B: AirSeal® Pneumoperitoneum and Moderate Blockade; Arm 3A: Conventional Pneumoperitoneum and Deep Blockade; Arm 3B: AirSeal® Pneumoperitoneum and Deep Blockade

SUMMARY:
The investigators are testing the hypothesis that lower pressure pneumoperitoneum during laparoscopic large bowel surgery protects the bowel from postoperative ileus and bowel dysfunction leading to faster recovery and discharge from the hospital. Our study will focus on the effects of high or low intraperitoneal pressure as well as pressure variations on the course of postoperative ileus, time to hospital discharge, and postoperative gastrointestinal dysfunction in adult patients undergoing laparoscopic large bowel resection (i.e., sigmoidectomy and right colectomy). A randomized parallel group study will be conducted involving 5 arms of surgical patients to test whether differences on postoperative ileus outcome parameters occur between high (15 mm Hg) and low pressure pneumoperitoneum (8-12 mm Hg), as well as whether there are differences between the 2 insufflation devices that provide constant or variable intrabdominal pressure throughout the laparoscopic surgery. For high pressure pneumoperitoneum, either neostigmine or sugammadex are used for reversal of moderate neuromuscular blockade. For low pressure pneumoperitoneum, sugammadex is used for reversal of deep neuromuscular blockade. The investigators plan to use 2 types of gas insufflation devices, one of which will provide a relatively stable pressure level throughout surgery (AirSeal® device), and the second one will provide a more variable pressure (Olympus standard insufflation device). Using both pressure modalities, the investigators will study the effects of different pressure characteristics on the course of postoperative ileus, duration of in-hospital treatment, pain level, and the stability of hemodynamic and respiratory parameters during surgery. Changes in intrabdominal pressure during the surgery will be monitored and recorded using a custom software for later analysis of fluctuations in pressure to relate them to outcomes. Other parameters will be obtained from EPIC (IHIS) medical charts. In addition, clinical data on postoperative ileus will be correlated with experimental outcomes from in vitro exploratory studies done using human samples of peritoneal lavage fluid, serum, and a small portion of the surgically removed bowel from each patient (that is otherwise discarded). A panel of inflammatory markers will be analyzed and biochemical, imaging, histological, immunochemical, molecular signaling, and glial activation studies will be done to evaluate the potential mechanisms of dysfunction associated with postoperative ileus.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients > 18 years old of both sexes who consent to participate in the study and do not have any of the exclusion criteria.
2. Patients undergoing laparoscopic right hemicolectomy to remove tumors.
3. Patients undergoing sigmoid resection to remove polyps, diverticula or tumors.

Exclusion Criteria:

1. History of inflammatory bowel disease.
2. History of intestinal ischemia.
3. History of intestinal adhesions and adhesive disease.
4. Patients with a history of bowel resection or major abdominal surgery in the past. Appendectomies and hernia repairs are not considered exclusion criteria.
5. Patients having epidural catheters placed for postoperative pain control for the study period. Intrathecal morphine injections for postoperative pain control will not exclude the patients from the study.
6. Significant acid-base and electrolyte imbalance before surgery as determined by the study personnel at the screening stage.
7. Allergy to or contraindications to rocuronium, or sugammadex.
8. Patients affected by medical conditions or receiving drugs that may prolong or shorten the duration of rocuronium effect (i.e. aminoglycosides, magnesium).
9. Significant comorbid conditions as determined by the study personnel at the screening stage.
10. Patients receiving any drugs that may significantly alter the picture of postoperative ileus (determined by the investigators) will be excluded from the study.
11. Prisoners and pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Length of time (hours) of postoperative gastrointestinal tract (GIT) function recovery | Up to 30 days after surgery. From "end of surgery" to "readiness for hospital discharge", i.e., physician discharge order (assessed up to 30 days after surgery).
  "Time from end of surgery to readiness for discharge" is used as a quantitative measure of postoperative gastrointestinal tract (GIT) function recovery and hence the length of postoperative ileus, and is an outcome used universally to estimate recovery of GIT function. The decision to discharge the patient ('time to discharge after surgery') by the physician is based on both the time of first spontaneous bowel movement after surgery (or flatus) and ability to tolerate a solid meal without vomiting/nausea. This parameter (time to discharge) can be measured reliably in every patient and in all 125 patients planned for enrollment in the study, increasing our chances of being able to detect differences between high and low pressure pneumoperitoneum.
Number of participants with postoperative ileus | Up to 4 days after surgery. From the "end of surgery" to Postoperative Day 4.
  Postoperative diagnosis of ileus by Day 4 after surgery (as defined by Vather et al. 2013). Reference: Defining Postoperative ileus: results of a systemic review and global survey. Journal of GI surgery, 2013. 17(5):p962-972.

SECONDARY OUTCOMES:
Number of participants with delayed postoperative ileus | Up to 5 days after surgery. From the "end of Surgery" to 5 days post-surgery as defined by Vather et al. (2013).
  This is calculated as the percent of subjects with postoperative gastrointestinal dysfunction (POGD) ≥5 days defined as subjects unable to tolerate solid foods, take anything by mouth, or requiring insertion or reinsertion of nasogastric tube at or after 5 days post-surgery
Time the participants will need to recover oral tolerance after surgery | Up to 30 days after surgery. From the "end of surgery" to first tolerated solid meal (assessed up to 30 days after surgery).
  Time to first tolerated solid meal: defined as the time each participant will take to eat the first solid meal without experiencing clinically significant nausea and/or vomiting for 1 calendar day after the meal.
Time the participants will need to have their first bowel movement occurrence after surgery | Up to 30 days after surgery. From the "end of surgery" to first spontaneous bowel movement (assessed up to 30 days after surgery).
  The time participants will take to experience their first bowel movement occurrence after surgery. This outcome is one of the main clinical signs of postoperative gastrointestinal function recovery.
Time the participants will need to have their first flatus after surgery | Up to 30 days after surgery. From the "end of surgery" to first spontaneous flatus (assessed up to 30 days after surgery).
  The time participants will take to experience their first flatus occurrence after surgery. This outcome is one of the main clinical signs of postoperative gastrointestinal function recovery.
Number of participants with postoperative ileus as only complication | Up to 30 days after surgery. From "end of surgery" to "readiness for hospital discharge", i.e., physician discharge order (assessed up to 30 days after surgery).
  Investigators will report the incidence of postoperative ileus as the only postoperative complication (i.e. isolated postoperative ileus without any other concomitant complication) which may offer significant information about the impact of postoperative ileus on delayed gastrointestinal tract recovery and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Fedias L Christofi, Ph.D., AGAF, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Tzagournis Medical Research Facility, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No